CLINICAL TRIAL: NCT07011485
Title: A Triple-Blind, Randomized, Efficacy and Tolerability Comparison Study of PDFE-2304 Topical Solution Versus Minoxidil 5% Topical Solution for the Treatment of Androgenic Alopecia (AGA).
Brief Title: A Safety and Efficacy Study of PDFE-2304 Topical Solution for the Treatment of Androgenic Alopecia.
Acronym: NEOPILI-2A
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PDFE Pharma Innovations FZCO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PDFE-CL-24-001
Record Dates: First submitted 2025-05-14; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Alopecia, Androgenetic; Baldness; Androgenetic Alopecia (AGA)
Keywords: Double Blind; Randomized; Efficacy; Tolerability; Comparison; Treatment
MeSH Terms: conditions — Alopecia | interventions — Minoxidil; Solutions

STUDY DESIGN:
Intervention Model Description: Parallel-group (2:1)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PDFE-2304 Topical Solution (Experimental): Approximately one mL dose applied onto a pre-specified scalp area twice daily for 16 weeks.
  Interventions: Drug: PDFE-2304 Topical Solution
- Minoxidil 5% Topical Solution (Active Comparator): Approximately one mL dose applied onto a pre-specified scalp area twice daily for 16 weeks.
  Interventions: Drug: Minoxidil 5% Topical Solution

INTERVENTIONS:
Drug: Minoxidil 5% Topical Solution — Approximately one mL dose applied onto a pre-specified scalp area twice daily for 16 weeks.
  Arms: Minoxidil 5% Topical Solution
Drug: PDFE-2304 Topical Solution — Approximately one mL dose applied onto a pre-specified scalp area twice daily for 16 weeks.
  Arms: PDFE-2304 Topical Solution

SUMMARY:
This study will evaluate the safety and efficacy of PDFE-2304 compared with Minoxidil 5% in men with androgenic alopecia (AGA).

ELIGIBILITY:
Inclusion Criteria -

* Men who have a presentation of androgenetic alopecia (Norwood II - V).
* Age between 18 to 60 years of age (both inclusive).
* Have no abnormal findings during physical examination.
* Able to comply with the study procedures in the opinion of the PI/CI.
* Able to give written consent for participation in the study.

Exclusion Criteria -

* Known hypersensitivity or idiosyncratic reaction to the API´s.
* Clinical diagnosis of non-AGA forms of alopecia.
* History of hair transplants.
* Subject having dyed or bleached hair 12 months prior to study start.
* Use of any topical product in the target region in the last 6 months.
* A medical history of receiving chemotherapy/cytotoxic agents.
* Uncontrolled hypertension.
* Any dermatological disorders (eczema, psoriasis, sun damage, skin cancer).
* Hormonal diseases such as thyroid disorders or diabetes.
* Liver and kidney disease.
* Smokers.
* Drug or alcohol abuse within 12 months.
* No written consent.
* The receipt of an investigational product or participation in a drug research study within a period of 90 days prior to the first dose of study drug.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2025-08-14 (Estimated); Study Completion 2025-09-17 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Target Area Hair Count (TAHC) | Baseline, Week 16 (Day 112)
  TAHC is measured using digital imaging analysis and is reported in terminal hairs/centimeters squared (cm^2). A positive change from Baseline indicates improvement (increase in the number of terminal hairs) and a negative change from Baseline indicates worsening (decrease in the number of terminal hairs).

SECONDARY OUTCOMES:
Percentage of Participants in Each Response Category of the Subject Self-Assessment in Alopecia (SSA) Score | Week 16 (Day 112)
  The SSA score measures scalp hair growth. Using a 7-point scale, participants will answer the Question: "Since the start of the study, the amount of my hair has?": Greatly Increased, Moderately Increased, Slightly Increased, Remained the Same, Slightly Decreased, Moderately Decreased or Greatly Decreased. The percentage of participants in each response category will be presented.
Percentage of Participants in Each Response Category of the Investigator Global Assessment (IGA) Score | Week 16 (Day 112)
  The investigator will compare the participant's scalp hair growth at Week 16 (Day 112) to a photograph of the scalp taken at Baseline and using the 7-point IGA score, the investigator will answer the question: "Since the start of the study, the amount of the subject's hair has?": Greatly Increased, Moderately Increased, Slightly Increased, Remained the Same, Slightly Decreased, Moderately Decreased or Greatly Decreased. The percentage of participants in each response category is presented.
Change From Baseline in Target Area Hair Width (TAHW) | Baseline, Week 16 (Day 112)
  Digital imaging analysis will be used to measure TAHW in millimeters/centimeters squared (mm/cm^2). The diameters of all terminal hairs (individual hairs ≥ 30 microns in width) in the target area will be summed and reported together. A positive change from Baseline indicates improvement (increase in the diameter of terminal hairs) and a negative change from Baseline indicates worsening (decrease in the diameter of terminal hairs).
Change From Baseline in Target Area Hair Darkness (TAHD) | Baseline, Week 16 (Day 112)
  Digital imaging analysis will be used to measure TAHD. The darkness of all terminal hairs (individual hairs ≥ 30 microns in width) in the target area will be summed and divided by total number of terminal hairs in the same target area and will be reported as intensity units. A positive change from Baseline indicates improvement (increase in the darkness of terminal hairs) and a negative change from Baseline indicates worsening (decrease in the darkness of terminal hairs).
Percentage of Participants in Each Response Category of the Global Panel Review (GPR) Score | Week 16 (Day 112)
  At the completion of the study, 3 independent dermatologists using the 7-point GPR score compared photographs of the participant's scalp hair growth at Week 16 (Day 112) to Baseline will answer the question: "Compared with the baseline image, the amount of the subject's hair has?": Greatly Increased, Moderately Increased, Slightly Increased, Remained the Same, Slightly Decreased, Moderately Decreased or Greatly Decreased. The percentage of participants in each response category will be presented.
Adverse Events | Baseline, Week 16 (Day 112)
  Any undesirable experience associated with the treatment or the comparator in a study participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Koppal Institute of Medical Sciences, Koppal, Karnataka, India

IPD SHARING:
Plan to Share IPD: No
Legal and Regulatory Barriers